CLINICAL TRIAL: NCT05286671
Title: Evaluation of Perioperative Management of Curative Anticoagulants in the Geriatric Perioperative Unit in Patient Hospitalized for Femoral Neck Fracture.
Acronym: ANTICOGER
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2022/CC-01
Record Dates: First submitted 2022-02-18; First posted 2022-03-18 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-03

CONDITIONS: Anticoagulants; Circulating, Hemorrhagic Disorder; Femoral Neck Fractures
Keywords: older patients; anticoagulant; femoral neck fractures; clinical pharmacy service
MeSH Terms: conditions — Hemorrhagic Disorders; Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pilot study to evaluate the management of curative anticoagulant prescriptions pre- and postoperatively in elderly patients hospitalized for femoral neck fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patient 75 years or older
* Hospitalized in the geriatric perioperative unit for a femoral neck fracture between 18/11/2019 and 30/06/2021
* Treated with a curative anticoagulant at entry
* Patient enrolled in or receiving a social security plan

Exclusion Criteria:

* Orthopedic patient housed in the geriatric perioperative unit
* Patient who objected to the use of their data

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients aged 75 years and older, hospitalized in the geriatric perioperative unit from November 18, 2019 to June 30, 2021, for a hip fracture and with curative anticoagulant therapy prescription at entry.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Rate of compliance with the recommendations for direct oral anticoagulants (DOAC).. | Day 0
  Rate of compliance with the french working group on perioperative haemostasis (GIHP) recommendations for DOACrecommendations for DOA.
Rate of compliance with the recommendations for vitamin K antagonists (VKA). | Day 0
  Rate of compliance with the french health authority (HAS) recommendations for VKA

SECONDARY OUTCOMES:
Number of pharmaceutical interventions | Day 0
  Number of pharmaceutical interventions regarding anticoagulant prescriptions
description of pharmaceutical interventions | Day 0
  description of pharmaceutical interventions
Evaluation of the morbi-mortality | Day 0
  Mortality, re-hospitalizations at 30 days, characterization of bleeding complications, characterization of thrombotic complications
Description of the evolution of the plasma dosage of DOAC and the international normalized ratio (INR) and analysis of the operative delay | Day 0
  Value of preoperative DOAC plasma dosage, value of INR dosage pre- and post-op, analysis of the operative delay
description of the population | Day 0
  age, weight, height, body mass index, comorbidities

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No